CLINICAL TRIAL: NCT06394609
Title: Arthroscopic Bankart Repair Using Double Loaded Grand Knot Technique Versus Double Loaded Knotted Suture Anchor; Comparative Study
Brief Title: Comparison of Arthroscopic Bankart Repair Using Double Loaded Grand Knot Technique Versus Double Loaded Knotted Suture Anchor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Assistant Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-472-2018
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Arthroscopic Bankart Repair
Keywords: Arthroscopic Bankart Repair; double loaded Grand Knot Technique; Double loaded knotted suture Anchor; traumatic anterior shoulder instability

STUDY DESIGN:
Intervention Model Description: Patients with recurrent anterior glenohumeral subluxation or dislocation after an initial episode of traumatic anterior shoulder dislocation, a Bankart lesion confirmed by Magnetic resonance imaging (MRI) and arthroscopic examination. We would like to report the 12 months clinical outcomes of double loaded grand knot technique and knotted double loaded anchor used in traumatic anterior dislocations of the shoulder
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- double loaded knotted suture anchor (Experimental): arthroscopic bankart repair by using double loaded knotted suture anchor
  Interventions: Other: double loaded knotted suture anchor; Other: double grand knot

INTERVENTIONS:
Other: double loaded knotted suture anchor — arthroscopic bankart repair by using double loaded knotted suture anchor
Other: double grand knot — arthroscopic bankart repair by using double grand knot

SUMMARY:
Arthroscopic surgery is the preferred method to fix a Bankart lesion (tears in the labrum) and has better patient outcomes. It's important to assess any bone loss in the shoulder socket before surgery for a successful outcome. Using suture anchors to reattach the torn tissue is advantageous because it avoids going through the back of the shoulder. The article describes a specific technique for tying the sutures and anchor placement to minimize nerve and artery damage. Design of the suture anchor and how the suture is placed can affect its strength. Using two sutures per anchor (double-loaded) might be just as strong as using three anchors with one suture each (single-loaded), which is more common. This could save cost and bone but needs further study. The study proposes a new surgical technique using double-loaded anchors with more sutures to see if it offers similar strength while reducing implant use.

DETAILED DESCRIPTION:
Anatomical repair of the capsulolabral complex of the glenoid has become the gold- standard treatment for traumatic anterior shoulder instability associated with Bankart lesion.Arthroscopic technique results was better in postoperative functional outcome. (1) Specific findings in the history and the physical examination provide important clues to the presence of glenoid bone loss, and a careful preoperative evaluation to diagnose and quantify anterior glenoid deficiency is crucial for the success of surgical treatment. (2)

The use of suture anchors technique has the advantage of allowing the capsuloligamentous structures to be shifted superiorly and properly tensioned without the need to penetrate posteriorly. (3)

The grand knot is a double loop with an alternative half hitches 5 clock and 5 anticlockwise with total 30 hitches (big enough to hang on bony tunnel made by the guide wire). The anchors hanged over the posterior glenoid by pull out technique using number 2 proline introduced by the guide wire through the anterior portal. Skin exit will be 2 cm lateral and 5 cm inferior to postero-lateral corner of the acromion (safe zone) by which, the low postero-lateral portal will be 1.5 cm away from axillary nerve and 1.4 cm away from the posterior humeral circumflex artery to avoid any neurovascular injury. (4) Simple attention to potential variations in the origin and course of the axillary nerve and its relationship to the shoulder capsule and having a precise knowledge of ''safe zones'' during operations can enhance surgical outcomes. (5) Abrasion of the suture during intraoperative and postoperative cyclic loading may be an important cause of suture weakening and breakage. This situation may be made worse by angulation of the suture with respect to the anchor's axis (SA) and by the rotational orientation of the anchor's eyelet with respect to the plane of the suture (RA) (6) The use of double loaded suture anchors can provide biomechanical strength equivalent to that provided by the currently recommended and frequently used single-loaded 3- anchor constructs. The use of more suture anchors has negative implications for the biomechanical strength of the repair and compromises glenoid fixation and bone stock Using fewer anchors with more sutures per anchor may protect glenoid bone stock while achieving comparable biomechanical stability. (7) Arthroscopic double-loaded single-row repair using suture anchors containing two non- absorbable braided sutures in chronic anterior shoulder dislocation is reliable procedure with respect to recurrence rate, range of motion, and shoulder function. (8) The following study is aiming to assess the functional outcomes after arthroscopic bankart repair using double loaded grand knot technique that increase number of sutures which hypothetically provide better biomechanical strength in repairing capsule

-labral complex with reduced implants costs and compare it with using double loaded anchors in patients who will be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent anterior glenohumeral subluxation or dislocation after an initial episode of traumatic anterior shoulder dislocation, a Bankart lesion confirmed by arthroscopic examination and Magnetic resonance imaging (MRI)

Exclusion Criteria:

1. Significant bony pathology (bony bankart)
2. Poor quality capsule-labral tissue
3. Multi directional instability
4. Ligamentous laxity
5. ALPSA lesion
6. Hillsachs lesion more than 10 %

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Constant score | 12 months

SECONDARY OUTCOMES:
ASES Shoulder Score | 12 months
Rowe score | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rashwan AS, Amin AQ, Zawam SH, Soliman AM, El-Desouky M. Arthroscopic Bankart repair using trans-glenoid double-loaded grand knots versus double-loaded suture anchors; is there a difference? a randomized controlled study. BMC Musculoskelet Disord. 2025 Mar 21;26(1):280. doi: 10.1186/s12891-025-08477-3. PMID 40114187